CLINICAL TRIAL: NCT04574453
Title: A Randomized, Open Label, Paralel Goup Study To Assess With A Non- Inferiority Hypothesis The Efficacy And Safety Of The Medical Device Iracross (Crosslinked 2% Hyaluronic Acid) Versus The Medical Device Iraline (Linear 2% Hyaluronic Acid), Administered Intra-Articular To Patients With Knee Osteoarthritis
Brief Title: Study To Assess The Efficacy And Safety Of The Medical Device Iracross Versus Iraline Administered Intra-Articular To Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.A. Istituto Ricerche Applicate S.p.A. (Network)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPIRA/0519/MD
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, open label, multicentre study with two parallel groups of patients and a non-inferiority hypothesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iracross (Experimental): 1 course of IRACROSS (crosslinked 2% Hyaluronic Acid) at baseline, consisting of a mono-dose intra-articular administration (2ml).
  Interventions: Device: Iracross
- Iraline (Active Comparator): 1 course of IRALINE (linear 2% Hyaluronic Acid); each course consists of 3-5 intra-articular administrations (2ml) at weekly intervals (from week 1 to 3, 4 or 5, depending on each patient's need)
  Interventions: Device: Iraline

INTERVENTIONS:
Device: Iracross — Administration of max 2ml of Iracross at first visit
  Arms: Iracross
Device: Iraline — Administration of maximum 2 ml of Iraline at visit 1 to visit 3, 4 and 5 depending of suject's need
  Arms: Iraline

SUMMARY:
Comparison with a non-inferiority design at 12 and 24 weeks on a larger scale is real to objectively evaluate the composite measurement of ROM, pain and basic activities like walking or performing daily activities (QoL) in a population with a large coverage of age and levels of physical activity (from no physical activity history to athletes).

DETAILED DESCRIPTION:
After giving their consent, subjects will undergo a screening visit to determine eligibility for study entry. After randomization, subjects will have administered medical device Iracross or Iraline. For subjects allocated to Iracross, medical device will be administered only at first visit and for subjects allocated to Iraline, medical device will be administered at visit 1, visit,2, visit 3 and optional for visit 4 and visit 5.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 40 and 80 years
2. Symptomatic knee osteoarthritis as defined by the American College of Rheumatology (ACR) criteria; (for subjects with OA at both knees, the most painful one will be included in the study only, respecting KL grade II or III);
3. Ambulant without assistance;
4. Kellgren-Lawrence grade II or III on X-ray performed at maximum 6 months before screening;
5. VAS knee pain ≥40 at screening and 30 days before;
6. At least 30 days before screening oral/parenteral corticosteroid or NSAIDs (10 mg prednisone) administration.
7. Signed Informed consent

Exclusion Criteria:

1. Unstable knee;
2. Varus or valgus ≥ 15 degrees;
3. Active malignancy;
4. Knee trauma or lose body parts 1 year before screening;
5. Rheumatoid Arthritis, avascular necrosis, fibromyalgia;
6. Use of potent analgesics 15 days (different from ≤ 10 mg prednisone);
7. Intra-articular HA or corticosteroid injection within 6 months before screening;
8. Arthroscopic or knee open surgery within 12 months before screening;
9. Body Mass Index (BMI) ≥ 40 kg/m2;
10. Active infection around the injection site;
11. Use of anticoagulants or history of thrombocytopenia;
12. Concomitant use of disease-modifying antirheumatic drugs (DMARDs), anaesthetics;
13. Known sensitivity to HA or DVS;
14. Pregnancy, breast feeding.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Change in Range Of Motion and Visual Analogue Scale | 180 days
  Change in ROM and VAS for pain (at rest), at 180 (± 4 days) days

SECONDARY OUTCOMES:
Physician Efficacy Global Evaluation | 180 days
  Score of Physician Efficacy Global Evaluation at final visit. Minimum value is4-poor efficacy and maximum value is 1- very good efficacy
Visual Analogue Scale Evaluation | 180 days
  VAS for pain (on moving and on pressing). Minimum score is 0 and it means no pain. Maximum score is 100 and represents the maximum pain that patient can suffer.
Knee injury and Osteoarthritis Outcome Score | 180 days
  Changes in KOOS score from first visit to final visit. The min value is 0 and the max value 100, were the min value represents no problem and max value represents extreme problems
NSAID consumption | 180 days
  Incidence of NSAID consumption from first visit to final visit

OTHER OUTCOMES:
AE, SAE, ADE, SADE, DD incidence. | 180 days
  To investigate the overall safety and tolerability of the two medical devices during the by overall study period.
Physician Global Tolerability | 180 days
  Percentage of patients with "excellent" evaluations in the Physician Global Tolerability Evaluation

CONTACTS AND LOCATIONS:
Overall Officials: George Puenea, Principal Investigator — Fizio Center
Locations (1):
- Fizio Center, Timișoara, Timiș County, Romania